CLINICAL TRIAL: NCT00230867
Title: A Multicenter, Placebo Controlled, Randomized, Double Blind, Subject Initiated Study of the Safety and Efficacy of a Single Topical Iontophoretic Application of Acyclovir 5% Cream With an Open Label Conventional Therapy Treatment Arm, and a Blinded Evaluator, for the Treatment of Recurrent Herpes Labialis
Brief Title: Iontophoretic Application of Acyclovir Cream to Treat Recurrent Herpes Labialis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Transport Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPI-203
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2006-06

CONDITIONS: Herpes Labialis
Keywords: herpes labialis; cold sore; acyclovir; iontophoresis; topical
MeSH Terms: conditions — Herpes Labialis

INTERVENTIONS:
Device: iontophoretic acyclovir

SUMMARY:
Currently approved drugs for the treatment of herpes labialis (cold sores) exhibit low levels of efficacy due to the limited ability of the drugs to penetrate the skin to the site where the herpes virus is replicating. Iontophoresis uses electric current to enhance the delivery of drugs through the skin. This trial is testing a new iontophoretic device for the delivery of acyclovir cream to treat cold sores.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of iontophoretically-applied acyclovir 5% cream for the treatment of herpes simplex labialis lesions including an open label arm using Zovirax (acyclovir) Cream 5% as per standard of care in the same patient population. Subjects who meet the eligibility requirements at the screening/randomization visit will be randomized in a 1:1:1 ratio to one of the three treatment groups. After being enrolled and randomized into the study, subjects will be sent home with a locked kit containing the iontophoretic device with either active or placebo cream or a locked kit containing Zovirax Cream 5%. At first signs and/or symptoms of a recurrent herpetic episode (Stage 0 or 1, prodromal or erythema), the lesion will be confirmed by telephone interview with the subject, and upon confirmation of the lesion, the subject will be given the combination to the locked kit and instructed to begin treatment immediately, thereby initiating the Treatment Phase of the study. Subjects will be followed for at least 5 consecutive days post-treatment up until a maximum of 10 consecutive days post-treatment, until the herpes lesion is healed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject 18-75 years of age
2. Female subject must be using a medically acceptable form of birth control during the study. Acceptable birth control measures are abstinence, oral contraceptive pills or patch, injectable contraception, barrier contraceptives (condom, diaphragm with spermicide), IUD, surgical (hysterectomy, tubal ligation), vasectomized partner, or natural post menopausal inability to conceive.
3. Subject must have a history of recurrent herpes labialis and report at least 3 recurrences during the preceding 12 months.
4. Subject must provide voluntary written informed consent to participate in this study.

Exclusion Criteria:

1. Subjects with a pacemaker, or a history of cardiac arrhythmias or conduction abnormalities. Any subject with a medically confirmed history of cardiac arrhythmia including sinus arrhythmia, premature beat, heart block, atrial fibrillation, atrial flutter and pulsus alternans is to be excluded from the study.
2. Any evidence of active malignancy, immunodeficient disease, or use of immunomodifying drugs (e.g., systemic steroids) within 30 days prior to enrollment. Subjects who have completed therapy and are considered unlikely to relapse or who have had surgery and do not have any evidence of disease, are eligible for the study.
3. Subjects using topical steroids on or near the face or systemic (oral, intravenous) steroids within 30 days of enrollment; use of inhaled steroids does not exclude a subject from the study.
4. History of allergic or adverse response to acyclovir, or any related anti-viral drug, or the cream base.
5. In females of childbearing potential, a positive urine pregnancy test at time of screening.
6. Subject is considered unreliable or unable to understand or follow the protocol directions or is unable to comprehend or satisfactorily use the measurement scales as determined by investigator or designee at screening.
7. Subject has abnormal skin conditions that occur in the area ordinarily affected by cold sores which might affect the normal course of cold sores (e.g., eczema, psoriasis, albinism, or chronic vesiculobullous disorders).
8. Subject is currently enrolled in another clinical trial or has used an investigational drug/device within 30 days of enrollment.
9. Subject has previously participated in the current study (TPI-203).
10. Subject has used an anti-viral medication in the preceding 30 days.
11. Subject requires chronic use of analgesics, pain medication or non-steroidal anti-inflammatory agents (NSAIDs). If a subject is unlikely to get through the treatment phase of the protocol without requiring the use of analgesia for a chronic condition, e.g. back pain, recurrent daily headaches, the subject should be excluded.
12. Subject has a recent history of renal dysfunction or serious hepatic disease. Renal dysfunction encompasses both acute and chronic renal failure, the former resulting from the sudden loss of the ability of the kidneys to excrete wastes, concentrate urine, and conserve electrolytes and the latter the gradual and progressive loss of these capabilities. Examples of serious hepatic disease would include alcoholic liver disease, chronic hepatitis, autoimmune hepatitis and a variety of inherited diseases. The underlying cause of a documented recent mild increase in liver enzymes should be considered when deciding whether or not to exclude such a subject.
13. Subject has a history of alcoholism or drug abuse within the preceding 12 months. A subject with a history of a pathological pattern of alcohol use that causes a serious impairment of social or occupational functioning should be excluded. Such subjects may exhibit symptoms of tolerance and withdrawal along with other behavioral symptoms.
14. Subject is institutionalized.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1800
Dates: Start 2005-04; Study Completion 2005-12

PRIMARY OUTCOMES:
Clinician assessed duration of the herpetic episode measured from time of treatment until lesion healed. Lesion assessments for a minimum of 5 consecutive days and a maximum of 10 consecutive days.

SECONDARY OUTCOMES:
Clinician assessed prevention of progression to a classical lesion
Clinician assessed duration of classical herpetic lesions.
Clinician assessed duration of the herpetic lesion (aborted lesions will be assigned a duration of lesion value of 0 for the purposes of the statistical analysis).
Clinician assessed duration of the herpetic lesion hard scab.
Examine the safety of iontophoretic application of acyclovir 5% cream.
All assessments for a minimum of 5 consecutive days and a maximum of 10 consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Hull, MD, Principal Investigator — University of Utah
Locations (26):
- United States (26):
  - Radiant Research Birmingham, Birmingham, Alabama
  - Radiant Research Phoenix Southeast, Chandler, Arizona
  - Radiant Research Phoenix, Phoenix, Arizona
  - Radiant Research Scottsdale, Scottsdale, Arizona
  - Radiant Research San Diego, San Diego, California
  - Radiant Research Santa Rosa, Santa Rosa, California
  - Radiant Research St. Petersburg, Pinellas Park, Florida
  - Radiant Research Stuart, Stuart, Florida
  - Radiant Research West Palm, West Palm Beach, Florida
  - Radiant Research Atlanta West, Atlanta, Georgia
  - Radiant Research Atlanta, Atlanta, Georgia
  - Radiant Research Boise, Boise, Idaho
  - Radiant Research Chicago, Chicago, Illinois
  - Radiant Research Minneapolis, Edina, Minnesota
  - Radiant Research St. Louis, St Louis, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Radiant Research Cincinnati, Cincinnati, Ohio
  - Pediatric Clinical Trials International, Columbus, Ohio
  - Radiant Research Philadelphia, Philadelphia, Pennsylvania
  - Radiant Research Greer, Greer, South Carolina
  - J & S Studies, Inc., Bryan, Texas
  - Radiant Research Dallas North, Dallas, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Univeristy of Utah Health Sciences, Salt Lake City, Utah
  - Dermatology & Laser Center NW, Bellingham, Washington
  - Radiant Research Tacoma, Lakewood, Washington

REFERENCES:
- See also: Sponsor company website — http://www.transportpharma.com